CLINICAL TRIAL: NCT03652467
Title: The Safety and Efficacy of Deferoxamine Combined With Conventional Transarterial Chemoembolization in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: The Safety and Efficacy of Deferoxamine for Treating Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinan Military General Hospital (Other)
Responsible Party: Principal Investigator, Li Min, Director, Jinan Military General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JNZY20181245
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Deferoxamine; Transarterial chemoembolization; Unresectable hepatocellular carcinoma
MeSH Terms: interventions — Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deferoxamine (Experimental): Patients are treated with deferoxamine and conventional TACE.
  Interventions: Drug: Deferoxamine and conventional TACE
- Conventional TACE (Active Comparator): Patients are treated with conventional TACE.
  Interventions: Drug: Conventional TACE

INTERVENTIONS:
Drug: Conventional TACE — Conventional chemoembolization drugs are injected through hepatic artery.
  Other Names: TACE
  Arms: Conventional TACE
Drug: Deferoxamine and conventional TACE — Deferoxamine is injected before conventional transarterial chemoembolization.
  Other Names: Deferoxamine & TACE
  Arms: Deferoxamine

SUMMARY:
To investigate the safety and efficacy of deferoxamine (DFO) combined with conventional transarterial chemoembolization (TACE) in patients with unresectable hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
DFO, an iron chelator, is considered as a potential drug to the treatment of HCC. Ferrum is an important transition metal for organisms and the liver plays a major role in its storage. However, in pathologic conditions, it will lead to hepatocyte injury through the free radicals generated by excess iron. In addition, excess iron accumulation in the liver increases toxic free iron, which is closely associated with hepatic inflammation, as well as the development and progression of HCC. Reduction of iron is likely an important therapeutic targets for treating HCC. Iron reduction therapy has been efficacious in both in animal HCC models and results of clinical studies also suggest potential efficacy for HCC. DFO chelates iron by forming a stable complex that prevents the iron from entering into further chemical reactions. The investigators assume that DFO, combined with TACE, may provide additional efficacy in patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* The participant must have histologically-confirmed, unresectable HCC
* At least 1 measurable lesion, and overall tumor lesions occupying < 50% of liver volume
* The participant has provided signed informed consent
* No known allergy to contrast media
* Not pregnant
* No vascular anatomy or bleeding that would preclude catheter placement or emboli injection

Exclusion Criteria:

* Patients receiving concurrent radiotherapy or immunotherapy.
* Patients who have received previous chemotherapy, biological agents, or radiotherapy.
* Prior transarterial chemoembolisation (TACE) or transarterial embolisation (TAE).
* Prior liver transplantation or liver resection.
* Current or recent (within 10 days of study start) use of full-dose anticoagulants for therapeutic purposes.
* Patients with high risk esophageal/gastric varices.
* The participant has central nervous system (CNS) metastases or carcinomatous meningitis
* The participant has poorly-controlled hypertension [in other words (ie), blood pressure in abnormal range despite medical management]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in Participants With Unresectable Hepatocellular Cancer | First dose to date of progressive disease or death due to any cause [every 3 cycles up to 36 months (1 cycle=2 weeks)]
  PFS is defined as the time from the first day of therapy to the first evidence of disease progression or death from any cause. As classified according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, disease progression is having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of a new lesion. Participants who are alive and without disease progression and participants who did not progress and are subsequently lost to follow-up are censored at the last objective tumor assessment.

SECONDARY OUTCOMES:
Time to Progression | First dose to date of PD [every 3 cycles up to 36 months (1 cycle=2 weeks)]
  The time from first day of therapy to the first date of objective evidence of progressive disease (PD) by Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD is defined as having at least a 20% increase in sum of longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of new lesion. Time to PD is censored at the date of death or study discontinuation.
Overall Survival | First dose to date of death up to 36 months
  Overall survival (OS) is the duration from first dose to death due to any cause. OS is censored at last contact date for participants who are alive at the end of follow-up period or lost to follow-up.
Percentage of Participants With Complete Response or Partial Response | First dose to date of objective progressive disease (PD) or death up to 36 months
  Objective response rate (ORR) is defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR). As classified according to Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria, CR is the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm) and normalization of tumor marker level of non-target lesions. PR is having at least a 30% decrease in sum of longest diameter of target lesions.
Duration of Response | Time of first response (CR, PR or Stable disease) to disease progression, or death due to any cause [every 3 cycles up to 36 months (1 cycle=2 weeks)]
  Duration of response is the interval from the date of initial documented response [complete response (CR) , partial response (PR) or Stable disease] to the first documented date of disease progression, initiation of other (or additional) antitumor therapy is first reported, or death due to any cause. As classified according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, CR is the disappearance of all target lesions, PR is having at least a 30% decrease in the sum of the longest diameter of target lesions, and stable disease is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease. Disease progression is having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of a new lesion. Data are censored for participants who did not progress or die.
Tumor Necrosis | Baseline to the end of the study (up to 3 years, 36 months)
  Tumor necrosis is quantified in liver lesions greater than 2 cm at Baseline. When MRI showed many cut surfaces for a single tumor, tumor size and the size of necrotic area is measured by accumulation of the serial sections containing the tumor. Lipiodol accumulation without contrast enhance in tumor after TACE is regarded as an indication of necrosis. Tumor necrosis is assessed at Baseline and 1-3 days prior to the next scheduled transarterial chemoembolisation (TACE) till disease progression. The extent of tumor necrosis is presented as the percentage of the tumor volume at Baseline.
Number of Participants With Iron Reduction of Liver | Baseline to the end of the study (up to 3 years, 36 months)
  The iron of liver will be measured by MRI, where R2* and QSM is applied to present the quantity of iron. Iron reduction is assessed at Baseline and 1-3 days prior to the next scheduled transarterial chemoembolisation. The test will be repeated 1 -3 days after the therapy. The reduction of liver iron will be calculated accordingly.
The Prognostic Value of Reduction of Liver Iron | Prior to TACE at baseline, 1 -3 days after the therapy
  The iron of liver will be measured by MRI, where R2* and QSM is applied to present the quantity of iron. All patients will undergo MRI before TACE, and the test will be repeated 1 -3 days after the therapy till disease progression. The reduction of liver iron will be calculated accordingly. Based on the measurements mentioned above, the prognostic value of reduction of liver iron will be analyzed.
Number of Participants With Drug-Related Treatment-Emergent Adverse Events | First dose to 36 months
  Data presented are the number of participants who experienced treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), Grade 3 or higher TEAEs, or adverse events (AEs) leading to discontinuation of treatment that are considered by the investigator to be related to ramucirumab. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.

CONTACTS AND LOCATIONS:
Locations (1):
- 960th hospital of PLA, Jinan, Shandong, China